CLINICAL TRIAL: NCT06380595
Title: Complex Endovascular Aortic Repair in Inflammatory and Infective Perivisceral Abdominal Aortic Aneurysms and Thoracoabdominal Aortic Aneurysms (CEVARII)
Brief Title: Complex EVAR in Inflammatory and Infective Abdominal and Thoracoabdominal Aortic Aneurysms
Acronym: CEVARII
Status: Enrolling by invitation | Type: Observational
Sponsor: CEVARII (Other)
Collaborators: University of Iowa (Other); University of Colorado, Denver (Other); University of Trieste (Other); University of Copenhagen (Other); University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Mel J. Sharafuddin, MD, FACS, FSIR, Clinical Professor of Surgery and Radiology, University of Colorado, Colorado Springs
Other Study IDs: 23 -1533
Record Dates: First submitted 2024-03-01; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Abdominal Aortic Aneurysm; Aneurysm, Infected; Aneurysm, Mycotic; Abdominal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm
Keywords: Infected; Mycotic; Inflammatory; Aortic Aneurysm; INAA; IAA; Infective Native; Complex endovascular aortic repair
MeSH Terms: conditions — Aneurysm, Infected; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infective Native Abdominal Aortic Aneurysms (INAA): Infective native aortic aneurysms (INAA) are rare but highly morbid conditions that pose unique diagnostic and therapeutic challenges to the vascular surgeon.
  Patients with confirmed NAA who were treated with complex endovascular techniques at participating centers will be included in the registry.
  Interventions: Procedure: Complex endovascular aortic repair (cEVAR)
- Inflammatory aortic aneurysms (IAA): Inflammatory aortic aneurysms (IAA) are rare but highly morbid conditions that pose unique diagnostic and therapeutic challenges to the vascular surgeon.
  Patients with confirmed IAA who were treated with complex endovascular techniques at participating centers will be included in the registry.
  Interventions: Procedure: Complex endovascular aortic repair (cEVAR)

INTERVENTIONS:
Procedure: Complex endovascular aortic repair (cEVAR) — Complex endovascular aortic repair (cEVAR) collectively refers to the use of fenestrated/branched EVAR (f/bEVAR) or other EVAR variations allowing alternative visceral incorporation approaches, such as laser or radiofrequency (RF) fenestration or parallel endografts (snorkel, periscope, chimney or sandwich EVAR) to enable repair of perivisceral AAA (pvAAA), thoracoabdominal aortic aneurysms (TAAA), and aortic arch aneurysms.

SUMMARY:
Complex endovascular aortic repair in inflammatory and infective perivisceral abdominal aortic aneurysms and thoracoabdominal aortic aneurysms (CEVARII) study is a collaborative international effort among vascular surgeons to establish a database on the global experience in the management of INAAs and IAAs. Ethical approval for the study was obtained from the Colorado Multiple Institutional Review Board (COMIRB) under protocol number 23-1533.

DETAILED DESCRIPTION:
Infective Native and Inflammatory Aortic Aneurysms (INAA & IAA) are rare, morbid conditions with unique challenges. INAA & IAA share clinical and imaging similarities but differ significantly in pathophysiology, management, and prognosis. Open surgical repair of INAA & IAA is technically challenging and associated with higher complications.

Complex endovascular aortic repair in inflammatory and infective perivisceral abdominal aortic aneurysms and thoracoabdominal aortic aneurysms (CEVARII) study is a collaborative international consortium effort among vascular surgeons to establish a database on the global experience in the management of INAAs and IAAs. CEVARII study is IRB approved with the number 23-1533.

Knowledge gained will help generate consensus on how to best manage patients with inflammatory and infective aortic aneurysms involving the visceral and thoracoabdominal aorta.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 18 years old with a diagnosis of inflammatory abdominal aortic aneurysm (IAA) or infective native aortic aneurysms (INAA), who have undergone complex endovascular aortic repair (cEVAR) are eligible for inclusion in this study.

Exclusion Criteria:

* Suboptimal documentation of clinical, laboratory, and imaging findings
* Presence of prosthetic material (endograft or open graft material)
* Prior open or endovascular aortic repair
* Findings suspicious of secondary aorto-enteric or -bronchial fistulas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of two separate cohorts: 1) inflammatory aortic aneurysms (IAA) and 2) infective native aortic aneurysms (INAA). Patients with confirmed IAA or INAA who were treated with complex endovascular techniques at participating centers will be included in the registry.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary Graft Patency | up to 36 months
  Defined as uninterrupted blood flow with no interventions. Follow-up timeframes - 1, 6, 12, 24, and 36 months
Bowel Ischemia | 30 days
  Bowel Ischemia requiring surgical resection/not resolving with medical therapy. Outcome measures include the number of Participants with bowel ischemia after surgery.
Presence of aortic aneurysm endoleak after surgery | up to 30 days
  The technical repair success is defined as the exclusion of the aneurysm without Type I/III endoleak, and with preservation of at least the Superior Mesenteric Artery or the Celiac Artery. Outcome measures include the number of participants with type I endoleak, and the number of participants with type III endoleak.
Aneurysm-related mortality (ARM) | up to 30 days
  Outcome measures include the number of participants who died 30 days after the procedure.
Conversion to Open Surgical Repair (OSR) | up to 30 days
  Outcome measures include the number of participants whose cases converted from endovascular aortic aneurysm repair to open surgical repair.
Aortic rupture | up to 30 days.
  Outcome measures include the number of participants who had aortic rupture.
Post-operative infection-related complication (IRC) | up to 24 months
  Outcome measures include the number of participants who had a new post-operative infection-related complication (IRC) in treated aortic segments or endograft, new IRC in contiguous aortic segments, or persistent sepsis.
The duration of preoperative, perioperative, and postoperative duration of anti-microbial or immunosuppressive pharmacologic therapies. | up to 36 months
  Duration of antibiotics (in days) prescribed for Infective aortic aneurysm patients before and after the surgery. Duration of immunosuppressive drugs (in days) for inflammatory aortic aneurysm patients before and after the surgery

SECONDARY OUTCOMES:
Assessment of Adverse Events (AEs) described in the protocol. | up to 36 months
  Follow-up timeframes - 1, 6, 12, 24, and 36 months
All Cause Mortality | 24 months
  Any death occurring during the study period, regardless of cause. Timeframes: 1 yeas and 2 years
Continued Aortic sac growth. | up to 24 months
  Outcome measures include the number of participants who had continued sac growth (> 0.5 mm/6 month) despite appropriate reinterventions.

CONTACTS AND LOCATIONS:
Overall Officials: MEL J Sharafuddin, MD, Principal Investigator — Memorial Hospital Central, University of Colorado Healthcare
Locations (1):
- University of Colorado Healthcare, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CEVARII research project information and updates — https://cevarii.com/
- See also: CEVARII research project sign up link for interested sites. — https://redcap.link/CEVARII